CLINICAL TRIAL: NCT03923920
Title: Screening for Systemic Amyloidosis Via the Ligamentum Flavum
Acronym: ALF
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mazen Hanna MD, Principle Investigator, The Cleveland Clinic
Other Study IDs: 18-1512
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Amyloid; Amyloidosis; Spinal Stenosis; Transthyretin Amyloidosis; Primary Amyloidosis of Light Chain Type
Keywords: Biopsy; Surgery; Screening
MeSH Terms: conditions — Alzheimer Disease; Amyloidosis; Spinal Stenosis; Amyloidosis, Hereditary, Transthyretin-Related; Immunoglobulin Light-chain Amyloidosis | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ligamentum flavum tissue (may contain surrounding tissue and subcutaneous fat)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Stenosis Biopsy: Biopsy of ligamentum flavum tissue during spinal stenosis surgery sent to pathology for amyloid-specific analysis
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — During clinically-scheduled spinal stenosis surgery, ligamentum flavum tissue (which may contain surrounding tissue and subcutaneous fat) that is removed during the procedure will be sent to pathology to be analyzed with amyloid-specific staining.

SUMMARY:
The investigators will prospectively evaluate for the presence of amyloid deposits in ligamentum flavum (yellow ligament) tissue samples obtained from patients undergoing spinal stenosis surgery. Patients who have tissue that stains positive for amyloid will be referred to an amyloidosis specialist.

DETAILED DESCRIPTION:
Similar to carpal tunnel syndrome, spinal stenosis is associated with systemic amyloidosis and presents earlier than cardiac amyloidosis symptoms - 21-45% of ATTR patients and case reports in AL patients. The investigators' recent study found that 10% of older patients undergoing carpal tunnel release surgery were positive for amyloidosis, with 20% of that group presenting with cardiac involvement. 70% of the amyloid-positive group had a history of spinal stenosis and 40% required surgical intervention. Surgical intervention for spinal stenosis could provide an opportunity to screen for amyloidosis through yellow ligament (ligamentum flavum) biopsy.

This study will look at the prevalence of amyloidosis in patients undergoing surgical intervention for non-congenital spinal stenosis and spondyloarthropathy. The investigators hypothesize that 10% of such patients will be positive for amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* Undergoing surgical intervention for non-congenital spinal stenosis and/or spondyloarthropathy
* Able to consent

Exclusion Criteria:

* History of congenital spinal stenosis or congenital spondyloarthropathy

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spinal stenosis surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of amyloidosis in older patients undergoing spinal stenosis surgery | Baseline to 30 days
  Incidence of amyloid deposits in removed ligamentum flavum tissue of older patients undergoing spinal stenosis surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mazen A Hanna, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sperry BW, Reyes BA, Ikram A, Donnelly JP, Phelan D, Jaber WA, Shapiro D, Evans PJ, Maschke S, Kilpatrick SE, Tan CD, Rodriguez ER, Monteiro C, Tang WHW, Kelly JW, Seitz WH Jr, Hanna M. Tenosynovial and Cardiac Amyloidosis in Patients Undergoing Carpal Tunnel Release. J Am Coll Cardiol. 2018 Oct 23;72(17):2040-2050. doi: 10.1016/j.jacc.2018.07.092. PMID 30336828
- [Background] Yanagisawa A, Ueda M, Sueyoshi T, Okada T, Fujimoto T, Ogi Y, Kitagawa K, Tasaki M, Misumi Y, Oshima T, Jono H, Obayashi K, Hirakawa K, Uchida H, Westermark P, Ando Y, Mizuta H. Amyloid deposits derived from transthyretin in the ligamentum flavum as related to lumbar spinal canal stenosis. Mod Pathol. 2015 Feb;28(2):201-7. doi: 10.1038/modpathol.2014.102. Epub 2014 Sep 5. PMID 25189643
- [Background] Westermark P, Westermark GT, Suhr OB, Berg S. Transthyretin-derived amyloidosis: probably a common cause of lumbar spinal stenosis. Ups J Med Sci. 2014 Aug;119(3):223-8. doi: 10.3109/03009734.2014.895786. Epub 2014 Mar 12. PMID 24620715
- [Background] Sueyoshi T, Ueda M, Jono H, Irie H, Sei A, Ide J, Ando Y, Mizuta H. Wild-type transthyretin-derived amyloidosis in various ligaments and tendons. Hum Pathol. 2011 Sep;42(9):1259-64. doi: 10.1016/j.humpath.2010.11.017. Epub 2011 Feb 21. PMID 21334722
- [Background] Sekijima Y, Yazaki M, Ueda M, Koike H, Yamada M, Ando Y. First nationwide survey on systemic wild-type ATTR amyloidosis in Japan. Amyloid. 2018 Mar;25(1):8-10. doi: 10.1080/13506129.2017.1409706. Epub 2017 Nov 28. PMID 29182024
- [Background] M'bappe P, Grateau G. Osteo-articular manifestations of amyloidosis. Best Pract Res Clin Rheumatol. 2012 Aug;26(4):459-75. doi: 10.1016/j.berh.2012.07.003. PMID 23040361